CLINICAL TRIAL: NCT02030418
Title: The LEADLESS II IDE Study (Phase I): Safety and Effectiveness Trial for the Nanostim Leadless Pacemaker
Brief Title: The LEADLESS II IDE Study for the Nanostim Leadless Pacemaker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-02374
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Leadless Pacemaker (Experimental): VVIR pacing
  Interventions: Device: Leadless Pacemaker

INTERVENTIONS:
Device: Leadless Pacemaker — Patients will undergo an attempted leadless pacemaker implant

SUMMARY:
Prospective, non-randomized, single-arm, international multicenter, clinical safety and effectiveness of a leadless pacemaker system in patients who are indicated for a VVIR pacemaker.

Following completion of enrollments in the IDE, patients will continue to be enrolled in the continued access phase of the study under the same protocol.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of the leadless pacemaker system in treating patients with a slow heart rate or irregular heartbeats. The Nanostim leadless pacemaker provides bradycardia pacing as a pulse generator with built-in battery and electrodes, for permanent implantation in the right ventricle. As a leadless pacemaker, it does not need a connector, pacing lead, or pulse generator pocket, but it has the same operating principles as a conventional pacemaker.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have one of the clinical indications before device implant in adherence with Medicare, ACC/AHA/HRS/ESC single chamber pacing guidelines including:

   * Chronic and/or permanent atrial fibrillation with 2 or 3° AV or bifascicular bundle branch block (BBB block), including slow ventricular rates (with or without medication) associated with atrial fibrillation; or
   * Normal sinus rhythm with 2 or 3° AV or BBB block and a low level of physical activity or short expected lifespan (but at least one year); or
   * Sinus bradycardia with infrequent pauses or unexplained syncope with EP findings; and
2. Subject ≥18 years of age; and
3. Subject has life expectancy of at least one year; and
4. Subject is not enrolled in another clinical investigation; and
5. Subject is willing to comply with clinical investigation procedures and agrees to return for all required follow-up visits, tests, and exams; and
6. Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the IRB; and
7. Subject is not pregnant and does not plan to get pregnant during the course of the study.

Exclusion Criteria:

1. Subject has pacemaker syndrome, has retrograde VA conduction or suffers a drop in arterial blood pressure with the onset of ventricular pacing; or
2. Subject is allergic or hypersensitive to <1 mg of dexamethasone sodium phosphate; or
3. Subject has a mechanical tricuspid valve prosthesis; or
4. Subject has a pre-existing endocardial pacing or defibrillation leads; or
5. Subject has current implantation of either conventional or subcutaneous implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT); or
6. Subject has an implanted vena cava filter; or
7. Subject has evidence of thrombosis in one of the veins used for access during the procedure; or
8. Subject has an implanted leadless cardiac pacemaker; or
9. Subject had recent cardiovascular or peripheral vascular surgery within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivik Reddy, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (59):
- United States (50):
  - University Hospital - Univ. of Alabama at Birmingham, Birmingham, Alabama
  - Heart Center Research, LLC., Huntsville, Alabama
  - Scripps Health, La Jolla, California
  - USC University Hospital, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - Premier Cardiology, Inc, Newport Beach, California
  - Huntington Memorial Hospital, Pasadena, California
  - Sequoia Hospital, Redwood City, California
  - Mercy Medical Group - Cardiology, Sacramento, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Naples Community Hospital, Naples, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health, Orlando, Florida
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - University of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Sparrow Research, Lansing, Michigan
  - Munson Medical Center, Traverse, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Cardiac Arrhythmia and Pacemaker Center, Roslyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Medical Group HeartCare, Greensboro, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - Clinical Tex Research, LLC, Amarillo, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Intermountain Heart Rhythm Specialists, Murray, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Aurora Medical Group, Milwaukee, Wisconsin
- Australia (3):
  - The Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver General Hospital (U of BC), Vancouver, British Columbia
  - Kinsgston General Hospital, Kingston, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
  - Institut de Cardiologie de Quebec (Hospital Laval), Québec

REFERENCES:
- [Derived] Reddy VY, Miller MA, Knops RE, Neuzil P, Defaye P, Jung W, Doshi R, Castellani M, Strickberger A, Mead RH, Doppalapudi H, Lakkireddy D, Bennett M, Sperzel J. Retrieval of the Leadless Cardiac Pacemaker: A Multicenter Experience. Circ Arrhythm Electrophysiol. 2016 Dec;9(12):e004626. doi: 10.1161/CIRCEP.116.004626. PMID 27932427
- [Derived] Reddy VY, Exner DV, Cantillon DJ, Doshi R, Bunch TJ, Tomassoni GF, Friedman PA, Estes NA 3rd, Ip J, Niazi I, Plunkitt K, Banker R, Porterfield J, Ip JE, Dukkipati SR; LEADLESS II Study Investigators. Percutaneous Implantation of an Entirely Intracardiac Leadless Pacemaker. N Engl J Med. 2015 Sep 17;373(12):1125-35. doi: 10.1056/NEJMoa1507192. Epub 2015 Aug 30. PMID 26321198

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Leadless Pacemaker
Started | 952
Successful Implants | 917
2-Week Visit | 904
6-Week Visit | 884
3-Month Visit | 869
6-Month Visit | 844
Completed | 808
Not Completed | 144
Not completed — Death | 78
Not completed — Missed 12-Month Visit | 9
Not completed — Withdrawn | 57

BASELINE CHARACTERISTICS:
Population: Enrolled Population (De Novo)
Arm/Group | Leadless Pacemaker
Number analyzed (Participants) | 952
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 359
  Male | 593
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36
  Not Hispanic or Latino | 913
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 22
  Black or African American | 61
  White or Caucasian | 862
  Other (Not Specified) | 4
  American Indian / Alaska Native | 3
Region of Enrollment [Number; unit: participants]
  Canada | 101
  United States | 827
  Australia | 24
Pacemaker Indication [Count of Participants; unit: Participants]
  Chronic AF with 2nd or 3rd Degree AV Block or Bundle Branch Block, including slow ventricular rates | 529
  Sinus Rhythm with 2nd or 3rd Degree AV Block or Byundle Branch Block | 96
  Sinus Bradycardia with Infrequent Pauses or Unexplained Syncope | 330
LV Ejection Fraction [Mean (Standard Deviation); unit: percentage] — Population: 850 patients reporting LV ejection fraction data
  percentage
    number analyzed (Participants) | 850
    (all) | 57.9 (8.1)
Congestive Heart Failure [Count of Participants; unit: Participants] | 149
NYHA Class [Number; unit: participants] — The NYHA Functional Classification is used to classify people with heart failure:
  I No limitation of physical activity. Ordinary activity does not cause undue fatigue, palpitation or shortness of breath.
  II Slight limitation of physical activity. Comfortable at rest. Ordinary activity results in fatigue, palpitation, shortness of breath or chest pain.
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV Symptoms of heart failure at rest. Any physical activity causes discomfort. Population: NYHA Class evaluated for patients with congestive heart failure
  participants
    Class I: number analyzed (Participants) | 149
    Class I | 34
    Class II: number analyzed (Participants) | 149
    Class II | 57
    Class III: number analyzed (Participants) | 149
    Class III | 21
    Not Done: number analyzed (Participants) | 149
    Not Done | 37
Hypertension [Number; unit: participants] — Population: 736 patients reporting hypertension
  participants
    Controlled with Medication(s): number analyzed (Participants) | 736
    Controlled with Medication(s) | 690
    Uncontrolled: number analyzed (Participants) | 736
    Uncontrolled | 45
    Controlled Without Medication(s): number analyzed (Participants) | 736
    Controlled Without Medication(s) | 1
Diabetes [Number; unit: participants] — Population: 242 patients reporting diabetes
  participants
    Type I: number analyzed (Participants) | 242
    Type I | 14
    Type II: number analyzed (Participants) | 242
    Type II | 228
Diabetes Current Status [Number; unit: participants] — Population: 242 patients reporting diabetes
  participants
    Controlled with Diet: number analyzed (Participants) | 242
    Controlled with Diet | 44
    Controlled with Medication(s): number analyzed (Participants) | 242
    Controlled with Medication(s) | 191
    Uncontrolled: number analyzed (Participants) | 242
    Uncontrolled | 7
Hyperlipidemia [Number; unit: participants] — Population: 615 patients reporting hyperlipidemia
  participants
    Hyperlipidemia Controlled with Diet: number analyzed (Participants) | 615
    Hyperlipidemia Controlled with Diet | 90
    Hyperlipidemia Controlled with Medication(s): number analyzed (Participants) | 615
    Hyperlipidemia Controlled with Medication(s) | 509
    Uncontrolled Hyperlipidemia: number analyzed (Participants) | 615
    Uncontrolled Hyperlipidemia | 16
Peripheral Vascular Disease [Number; unit: participants] | 113
Cardiac Pulmonary History [Number; unit: participants]
  Coronary Artery Disease | 334
  Myocardial Infarction | 127
  Unstable Angina | 25
  Prior PTCA / Stents / Atherectomy | 144
  Prior CABG | 129
Prior Ablation [Number; unit: participants]
  AV Nodal | 17
  AFib / Aflutter | 78
  VT | 2
  Mini Maze, Thorascope / LAA Ligation | 2
  SVT/AVNRT Ablation | 12
  Wolff-Parkinson-White Syndrome | 2
  Unkown | 1
Tricuspid Valve Disease [Number; unit: participants]
  Insufficiency / Prolapse / Regurgitation | 184
  Repair / Replacement | 7
Arrhythmia History [Number; unit: participants]
  Ventricular | 43
  Non-Ventricular / Supraventricular | 727
Medications [Number; unit: participants]
  Antiarrhythmics (Class I) | 18
  Antiarrhythmics (Class III) | 62
  Anticoagulants | 571
  Antiplatelets | 407
  ACE Inhibitors | 249
  Angiotensin Receptor Blockers | 167
  Beta Blockers | 357

OUTCOME MEASURES:

1. Primary Outcome: Complication-Free Rate
Description: Complication is any device-or-procedure related serious adverse event, or serious adverse device effect, including those that prevented initial implantation. Percentage of participants free from complications are reported
Time Frame: 6 months
Population: Analyses of the primary safety and effectiveness endpoints are performed on the Intent to treat (ITT) population. The ITT population is defined as subjects who meet enrollment criteria, provide signed informed consent, and who have an attempted implant of the LP. The study required a sample size of 300 evaluable subjects. The 300-subject primary analysis cohort is defined as the first 300 enrolled subjects sorted by implant date and sheath insertion time.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Leadless Pacemaker: Subjects who signed an approved informed consent form and had an attempted Nanostim implant, with no pre-existing implanted pacemaker at the time of consent
Arm/Group | Leadless Pacemaker
Number analyzed (Participants) | 300
percentage of participants | 93.3 [89.9 to 95.9]
Statistical Analysis 1: Comparison: Leadless Pacemaker; Test type: Superiority — The primary safety hypothesis is: H0: CFR ≤ 86% vs. H1: CFR > 86% Where CFR is the Complication Free Rate. The CFR is estimated as a binomial proportion and the 95% confidence interval (CI) of CFR is calculated using the Clopper-Pearson exact method. The null hypothesis is rejected at the 2.5% significance level if the lower bound of this CI exceeds the Performance Goal (PG) of 86%; p < 0.001, 1-sided exact test for binomial proporti; binomial proportion = 93.3, 95% CI 2-sided [89.9 to 95.9]

2. Primary Outcome: Pacing Thresholds and R-wave Amplitudes Within the Therapeutic Range
Description: Success Rate is percentage of subjects who have acceptable pacing threshold and sensing amplitudes, which are defined as pacing threshold <=2.0V at 0.4 ms pulse width and R-wave amplitude either =>5.0 mV at the 6 month visit or => value at implant.
Time Frame: 6 months
Population: Analysis of the primary effectiveness endpoints was performed on subjects in the Intent to treat (ITT) population with a successful Nanostim Leadless Pacemaker implanted. This number included 289 of the 300 (96.3%) subjects in the ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leadless Pacemaker
Number analyzed (Participants) | 289
percentage of participants | 93.4 [89.9 to 96.0]
Statistical Analysis 1: Comparison: Leadless Pacemaker; Test type: Superiority — The primary effectiveness hypothesis is: H0: Rate ≤ 85.0% vs. H1: Rate > 85.0% where Rate is the proportion of subjects experiencing success, and success is defined as: pacing threshold voltage ≤ 2.0 V at 0.4 ms at 6-month visit and sensed R-wave amplitude either ≥ 5.0 mV at the 6-month visit or ≥ value at implant; p < 0.001, 1-sided exact test for binomial proporti — The null hypothesis is rejected at the 2.5% significance level if the lower bound of the CI exceeds the Performance Goal (PG) of 85%; binomial proportion = 93.4, 95% CI 2-sided [89.9 to 96.0]

3. Secondary Outcome: Appropriate and Proportional Rate Response During Graded Exercise Testing
Description: Temperature-based rate response feature was evaluated to determine whether an appropriate and proportional rate response was achieved during maximal effort graded treadmill exercise testing protocol (CAEP). All capable subjects who have completed the 6-minute walk test (6MWT) were asked to perform a maximal effort CAEP exercise protocol to demonstrate an appropriate and proportional response of sensor-indicated rate in graded exercise tests.
  Data from subjects who have completed the 6MWT and have completed at least stage 3 of the CAEP exercise protocol, or 3.6 metabolic equivalent of task (METs), were included in the analysis.
Time Frame: 3-6 months
Population: Subjects within the enrolled population with a successful implant who completed the six-minute walk test and completed at least stage 3 of the CAEP.
Measure: Mean (95% Confidence Interval); unit: 1/(minutes*metabolic equivalent task)
Arm/Group | Leadless Pacemaker
Number analyzed (Participants) | 30
1/(minutes*metabolic equivalent task) | 0.83 [0.73 to 0.93]
Statistical Analysis 1: Comparison: Leadless Pacemaker; Test type: Other — The hypothesis is intended to test whether the mean slope is within 35% of 1. The hypothesis is stated as follows: H0: absolute value (Mean Slope - 100%) ≥ equivalence margin, equal to 35% H1: absolute value (Mean Slope - 100%) < equivalence margin, equal to 35% The calculation of slope for individual subjects in the CAEP exercise protocol is done by setting the y-intercept to zero; p = 0.001, two 1-sided test (TOST); Slope = 0.83, 95% CI 2-sided [0.73 to 0.93], Standard Deviation 0.27

ADVERSE EVENTS:
Time Frame: Mean follow-up of 44.2 months post-implant (median 40.9 months)
Description: Regular investigator assessment of adverse events reported on a case report form. Seriousness and device-or-procedure relatedness for all reported events were based on the adjudications from an independent clinical events committee.
Arm/Group | Leadless Pacemaker
All-Cause Mortality (participants affected / at risk) | 276/952
Serious Adverse Events (participants affected / at risk) | 436/952
Other Adverse Events (participants affected / at risk) | 236/952
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leadless Pacemaker (N=952)
Malignant Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12)
Premature Battery Depletion (Product Issues) | 176 (180)
Pneumonia (Infections and infestations) | 10 (10)
Dizziness (General disorders) | 5 (6)
Loss of Normal Device Function due to Component Malfunction (Product Issues) | 26 (26)
Hemothorax (Injury, poisoning and procedural complications) | 2 (2)
Peripheral Vascular Disease (Vascular disorders) | 2 (2)
Heart Failure (Cardiac disorders) | 43 (52)
Cardiac Perforation Resulting in Tamponade and Requiring Intervention (Injury, poisoning and procedural complications) | 10 (10)
Infection, Local at Access Site, or Systemic (Infections and infestations) | 19 (22)
Vascular Access Complication: Access Site Bleeding (Injury, poisoning and procedural complications) | 7 (7)
Myocardial Infarction (Cardiac disorders) | 18 (25)
Choledocholithiasis (Hepatobiliary disorders) | 1 (1)
Cardiac Arrhythmias (Cardiac disorders) | 21 (23)
Elective Device Replacement (Cardiac disorders) | 8 (8)
Angina Pectoris (Cardiac disorders) | 11 (16)
Rib and Vertebra Fracture (Injury, poisoning and procedural complications) | 1 (1)
Decreased Level of Consciousness (General disorders) | 1 (1)
Stroke (Nervous system disorders) | 18 (18)
Accidental Injury (Injury, poisoning and procedural complications) | 2 (2)
Fall (Social circumstances) | 5 (5)
Dyspnea (General disorders) | 12 (12)
Hematoma Formation, Including Retroperitoneal Hematoma/Hemorrahge (Injury, poisoning and procedural complications) | 4 (4)
Bacteremia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 9 (9)
Cardiac Perforation/Pericardial Effusion not Requiring Intervention (Injury, poisoning and procedural complications) | 3 (3)
Pericarditis (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Cardiac disorders) | 4 (4)
Device Dislodgement (Injury, poisoning and procedural complications) | 9 (9)
Left Leg Weakness During Implant Procedure (Injury, poisoning and procedural complications) | 1 (1)
Threshold Elevation Resulting in Second LP Implant (Injury, poisoning and procedural complications) | 1 (1)
Embolism (Vascular disorders) | 3 (3)
Cardiac Perforation Requiring Intervention (Injury, poisoning and procedural complications) | 2 (2)
Valve Damage (Injury, poisoning and procedural complications) | 7 (7)
Change in Mental Status Post Procedure (Psychiatric disorders) | 2 (2)
Intermittent Capture (Product Issues) | 1 (1)
Pericardial Effusion or Rub (Injury, poisoning and procedural complications) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Mechanical Trauma (Injury, poisoning and procedural complications) | 3 (4)
Syncope (General disorders) | 12 (16)
Terminal Heart Disease (Cardiac disorders) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 12 (12)
GI Bleeding (Gastrointestinal disorders) | 7 (10)
Urinary Retention (Renal and urinary disorders) | 3 (3)
Acute Renal Failure (Renal and urinary disorders) | 2 (2)
Hernia (General disorders) | 2 (2)
Celulitis (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Inability to Interrogate or Program due to Programmer or Device Malfunction (Product Issues) | 5 (5)
Pacemaker Syndrome (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 2 (2)
Fever- Unknown Etiology (Investigations) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1)
Change in Mental Status (General disorders) | 4 (4)
Peripheral Edema (Cardiac disorders) | 1 (1)
Aortic Stenosis (Cardiac disorders) | 2 (2)
Death, Unknown Cause (General disorders) | 5 (5)
Threshold Elevation (Product Issues) | 2 (2)
Dehydration (General disorders) | 2 (2)
Multi-System Organ Failure (General disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 4 (4)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1)
Vascular Access Complication: Pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Detached Docking Button (Product Issues) | 2 (2)
Colitis (Infections and infestations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Ventricular Ectopy (Product Issues) | 1 (1)
Access Site Bleeding Event (Injury, poisoning and procedural complications) | 1 (1)
Pre-Syncope (General disorders) | 1 (1)
Temporary Loss of Pacing and Sensing (Product Issues) | 1 (1)
RV Lead Dislodgement (Surgical and medical procedures) | 3 (3)
Reduction in Lvef (Cardiac disorders) | 1 (1)
Pneumothorax (Injury, poisoning and procedural complications) | 1 (1)
Threshold Elevation Resulting in Retrieval of LP (Injury, poisoning and procedural complications) | 5 (5)
Undifferentiated Shock (General disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Pocket Hematoma (Pm) (Injury, poisoning and procedural complications) | 3 (3)
Damage to Vessels (Injury, poisoning and procedural complications) | 1 (1)
Pneumonitis (Infections and infestations) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 7 (7)
Allergic Reaction to Vancomycin (Immune system disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Inadequate Fixation of The LP During Implant Resulting in Device Migration (Product Issues) | 5 (5)
Device Pocket Infection (Biv ICD) (Infections and infestations) | 1 (1)
Femoral-Popliteal Bypass Graft Occlusion (Vascular disorders) | 1 (1)
Thromboemboli (Vascular disorders) | 2 (2)
Asystole During Implant Procedure (Injury, poisoning and procedural complications) | 2 (2)
Intermittent Loss of Device Telemetry (Product Issues) | 1 (1)
Excessive Bleeding (Injury, poisoning and procedural complications) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Hypertension (Cardiac disorders) | 2 (2)
End Stage Renal Disease (Renal and urinary disorders) | 1 (1)
Vascular Access Complication: AV Fistula (Injury, poisoning and procedural complications) | 2 (2)
Chest Pain (General disorders) | 4 (4)
Failure to Capture/Loss of Capture (Product Issues) | 3 (3)
Seizure (Nervous system disorders) | 1 (1)
Leg Ischemia (Vascular disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Intracranial Hemorrhage (Nervous system disorders) | 2 (2)
Aortic Dissection (Vascular disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Weakness (General disorders) | 1 (1)
RV Pacing Induced Cardiomyopathy (Cardiac disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1)
Shoulder Dislocation (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (General disorders) | 1 (1)
Mechanical Trauma to His Bundle (Injury, poisoning and procedural complications) | 1 (1)
Contrast Induced Nephropathy (Injury, poisoning and procedural complications) | 1 (1)
Endocarditis of Prosthetic Valves (Infections and infestations) | 1 (1)
Hand Swelling (General disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Bell's Palsy (Nervous system disorders) | 1 (1)
Vertigo (General disorders) | 1 (1)
Tricuspid Valve Regurgitation (Cardiac disorders) | 1 (1)
Intermittent Complete Heart Block During Implant Procedure (Product Issues) | 1 (1)
Perclose System Malfunction (Injury, poisoning and procedural complications) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leadless Pacemaker (N=952)
Inadequate Fixation of The LP (Injury, poisoning and procedural complications) | 1 (1)
Dyspnea (Injury, poisoning and procedural complications) | 18 (20)
Premature Battery Depletion (Product Issues) | 43 (44)
Vascular Access Complication: Access Site Bleeding (Injury, poisoning and procedural complications) | 26 (26)
Reaction to Contrast (Injury, poisoning and procedural complications) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (General disorders) | 15 (15)
Pneumonia (Infections and infestations) | 2 (2)
Threshold Elevation (Injury, poisoning and procedural complications) | 9 (9)
Hypertension (Vascular disorders) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1)
Dizziness (General disorders) | 10 (11)
Dehydration (General disorders) | 2 (2)
Pain (General disorders) | 8 (9)
Chest Pain (General disorders) | 6 (6)
Accidental Injury (Injury, poisoning and procedural complications) | 3 (3)
Reaction to Sedation (Injury, poisoning and procedural complications) | 1 (1)
Unsuccessful LP Retrieval (Product Issues) | 2 (2)
Undersensing (Product Issues) | 3 (3)
Cardiac Arrhythmias (Cardiac disorders) | 20 (22)
Detached Docking Button (Product Issues) | 3 (3)
Pre-Syncope (General disorders) | 5 (5)
Hematoma Formation, Including Retroperitoneal Hematoma/Hemorrahge (General disorders) | 5 (5)
Angina Pectoris (Cardiac disorders) | 7 (7)
Heart Failure (Cardiac disorders) | 7 (7)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Tricuspid Valve Regurgitation (Injury, poisoning and procedural complications) | 2 (2)
Pacemaker Syndrome (Product Issues) | 6 (6)
RV Pacing Induced Cardiomyopathy (Cardiac disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Coughing With RV Pacing (Product Issues) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Exit Block (Cardiac disorders) | 1 (1)
Hypercalcemia (Investigations) | 1 (1)
Inability to Interrogate or Program due to Programmer or Device Malfunction (Product Issues) | 2 (2)
Infection, Local at Access Site, or Systemic (Infections and infestations) | 8 (8)
Loss of Normal Device Function due to Component Malfunction (Product Issues) | 13 (14)
Temporary Loss of Vision (Eye disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mild Skin Reaction to Pre-Procedural Prep (Skin and subcutaneous tissue disorders) | 1 (1)
Open Wound (Injury, poisoning and procedural complications) | 1 (1)
Hand Injury (Injury, poisoning and procedural complications) | 1 (1)
Nickel Allergy (Product Issues) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (2)
Mechanical Trauma (Injury, poisoning and procedural complications) | 2 (5)
Cardiac Perforation/Pericardial Effusion not Requiring Intervention (Cardiac disorders) | 2 (2)
Valve Damage (Cardiac disorders) | 1 (1)
Inability to Release Snare from Docking Button (Product Issues) | 2 (2)
High Impedance (Product Issues) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 2 (2)
Left Sided Numbness (Nervous system disorders) | 1 (1)
Helix Distortion (Product Issues) | 1 (1)
Migraines (General disorders) | 1 (1)
Failure to Capture/Loss of Capture (Product Issues) | 5 (5)
Palpitations (Cardiac disorders) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vascular Access Complication: Access Site Lymphatic Drainage (Injury, poisoning and procedural complications) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Access Site Bleeding Event (Injury, poisoning and procedural complications) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Memory Loss (Psychiatric disorders) | 1 (1)
Abscess of The Neck (Infections and infestations) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1)
Extra-Cardiac Pacing Stimulation (Product Issues) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Bruising (Blood and lymphatic system disorders) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Stasis Ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Anemia (General disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Thromboemboli (Injury, poisoning and procedural complications) | 1 (1)
Thrombophlebitis (Injury, poisoning and procedural complications) | 1 (1)
Intermittent Loss of Device Telemetry (Product Issues) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Essential Tremor (Nervous system disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Elevated Troponin (Investigations) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Vascular Access Complication: AV Fistula (Injury, poisoning and procedural complications) | 1 (1)
Contrast Extravasation at Groin Access Site (Injury, poisoning and procedural complications) | 1 (1)
Anesthesia Related Side Effect (General disorders) | 1 (1)
Interruption of Desired Pacemaker Function due to Electrical Interference (Product Issues) | 1 (1) — Either Electromyogenic or Electromagnetic
Chest Discomfort (General disorders) | 1 (1)
Elevated Inr (Investigations) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Uvulitis After Implant Procedure (Injury, poisoning and procedural complications) | 1 (1)
Tricuspid Regurgitation (Cardiac disorders) | 1 (1)
Pleural Effusions (Injury, poisoning and procedural complications) | 2 (2)
Spine Fracture (Injury, poisoning and procedural complications) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 2 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asystole During Implant Procedure (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Although the LEADLESS II Phase 1 study met the primary and secondary endpoints, the Nanostim LP device was not commercialized in the US and commercial sales in the EU were discontinued in 2016. The Nanostim LP device was redesigned into the Aveir VR LP device- evaluated in the LEADLESS II Phase 2 study (NCT04559945.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT02030418/Prot_SAP_000.pdf